CLINICAL TRIAL: NCT02330003
Title: A Randomized, Active-Comparator, Open-Label, Phase 1 Clinical Trial to Assess the Safety of the 'IL-YANG Inactivated Split Influenza Vaccine' and Fluarix Prefilled Syringe in Healthy Korean Male Volunteer
Brief Title: Phase 1 Study to Assess the Safety of Inactivated Split Influenza Vaccine and Control Vaccine in Korean Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Il-Yang Pharm. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IY_IFEZ_102
Record Dates: First submitted 2014-12-29; First posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: Influenza; Influenza vaccine; Split influenza vaccine; Seasonal influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IL-YANG PFS (Experimental): IL-YANG FLU Vaccine Prefilled Syringe INJ.
  Interventions: Biological: IL-YANG FLU Vaccine Prefilled Syringe INJ.
- TIV PFS (Active Comparator): Fluarix Prefilled Syringe
  Interventions: Biological: Fluarix Prefilled Syringe

INTERVENTIONS:
Biological: IL-YANG FLU Vaccine Prefilled Syringe INJ. — Second vaccination (only for the test group) of IL-YANG FLU Vaccine Prefilled Syringe INJ.0.5mL
  Arms: IL-YANG PFS
Biological: Fluarix Prefilled Syringe — Fluarix Prefilled Syringe 0.5mL
  Arms: TIV PFS

SUMMARY:
The purpose of this study to evaluate the safety of IL-YANG Inactivated Split Influenza Vaccine (IL-YANG FLU Vaccine Prefilled Syringe INJ.) in comparison with Fluarix Prefilled Syringe (inactivated split influenza vaccine) after single-dose intramuscular administration.

DETAILED DESCRIPTION:
This was a randomized, open-label, active-controlled clinical study. After providing voluntary written informed consent, subjects underwent protocol-specific assessments and tests within the 4 weeks prior to administration of the study vaccine, and those who met all of the inclusion/exclusion criteria were randomized sequentially to the test group or the comparator group according to the pre-generated randomization code. To investigate the safety of the study drug with a two-dose regimen in children, the test group received another dose 28 days after the first dose.

The investigator evaluated the safety and immunogenicity for each subject throughout the study. Safety assessments were performed 28 days after the first dose (Visit 4, End-of-Study Visit) for the comparator group receiving a single-dose regimen of Fluarix Prefilled Syringe, and for the test group receiving a two-dose regimen of the test drug, 28 days after the first dose (Visit 4) and 28 days after the second dose (Visit 6, End-of-Study Visit). Subjects were instructed to record any adverse event occurring after vaccination in the Patient Diary Card. For the immunogenicity assessment, an antibody titer test was performed prior to dosing at Visit 2 (baseline) and 28 days (Visit 4) after the first vaccination for both the test group and comparator group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between 20 and 55 years of age at screening
* Body weight of ≥ 55kg and within ±20% of ideal body weight (ideal body weight = (height cm - 100)*0.9) at screening
* Subjects with no congenital or chronic disease who were considered suitable for the study after screening assessments (investigator's opinion, medical history, physical examination, laboratory test, chest X-ray, and ECG) conducted within 28 days prior to vaccination
* Subjects who were given, and fully understood, the information about the study, made a voluntary decision, and provided written informed consent, to participate in the study and comply with all applicable study requirements

Exclusion Criteria:

* Subjects who have known or suspected infection with HAV, HBV, HCV, HIV or VDRL
* Subjects who have concurrent or a past history of immune deficiency disease
* Subject who had participated in blood donation within 1 week prior to vaccination, or are planning to participate in blood donation from Day 1 until Month 7 post-vaccination
* Subject with a history of Guillain-Barre syndrome
* Subject with hemophilia or thrombocytopenia, or being treated with an anticoagulant, who are at increased risk of serious bleeding during intramuscular injection
* Subjects who have concurrent or a past history of, malignant tumor of internal organ or blood vessels or skin metastasis
* Subjects with known allergy to a drug, food or latex, who had a history of anaphylaxis
* Subjects who had an acute fever with body temperature > 38.0 Cº within 72 hours prior to administration of the study vaccine or symptoms of suspected acute disease within 14 days prior to administration of the study vaccine
* Subjects who received another experimental drug or vaccine within 28 days before administration of the study vaccine or are planning to receive another experimental drug or vaccine during the study.
* Subjects who had previously received immunoglobulin or blood-derived products within the last 3 months prior to administration of the study vaccine, or are expecting to be treated with immunoglobulin or blood-derived products during the study
* Subjects who had received, or are scheduled to receive, systemic immunosuppressive therapy, radiation therapy or high-dose corticosteroid therapy within the last 6 months prior to administration of the study
* Subjects with a history of, or suspected, drug abuse based on subject interview and physical examination.
* Subjects with excessive consumption of caffeine and alcohol and excessive smoking
* Subject with a known allergy to eggs, chicken, or any components of the study vaccine
* Subjects who in the investigator's opinion, may not be suitable for vaccination or who may interfere with the objective assessment of the study outcomes.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Solicited local & general Adverse Event, Unsolicited Adverse Event | up to Day28(+7)
  Solicited local reaction: pain, tenderness, redness, swelling, Solicited general reactions: fever, nausea/vomiting, diarrhea, headache, fatigue, myalgia
Percentage of subjects achieving seroconversion and seroprotection for HI antibody after administration of the study vaccine | up to Day28(+7)
  Seroconversion: a pre-vaccination (Day 0) hemagglutination-inhibition (HI) antibody titer < 1:10 and a post-vaccination (Day 28) HI antibody titer ≥ 1: 40 (Case 1), or a pre-vaccination (Day 0) HI antibody titer ≥ 1:10 and a minimum four-fold rise in post-vaccination (Day 28) HI antibody titer (Case 2).
  Seroprotection: post-vaccination (Day 28) HI antibody titer ≥ 1:40

SECONDARY OUTCOMES:
Vital signs | up to Day28(+7)
Physical examination | up to Day28(+7)
ECG result | up to Day28(+7)
Clinical laboratory results | up to Day28(+7)
GMT of HI antibody titer before vaccination and after vaccination | up to Day28(+7)
  Geometric Mean Titer (GMT), as measured by pre-vaccination (Day 0) HI antibody titer and post-vaccination (vaccination + 28 days) HI antibody titer.
GMR of HI antibody titer before vaccination and after vaccination | up to Day28(+7)
  Geometric Mean Ratio (GMR), as measured by pre-vaccination (Day 0) HI antibody titer and post-vaccination (vaccination + 28 days) HI antibody titer
Percentage of subjects with a pre-vaccination (Day 0) HI antibody titer < 1:40, and a minimum four-fold rise in post-vaccination (Day 28) HI antibody titer | up to Day28(+7)

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, M.D,PhD, Principal Investigator — Severance Hospital, Yonsei University Health System